CLINICAL TRIAL: NCT07370064
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of Anti-CLL1-CD33-NKG2D Bicephali CAR-T Cells in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Clinical Study of Anti-CLL1-CD33-NKG2D Bicephali CAR-T for Relapsed/Refractory Acute Myeloid Leukemia
Acronym: AML CAR-T
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Principal Investigator, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL517-01; XYFY2025-KL517-01 (Other: The Affiliated Hospital oh Xuzhou Medical University)
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: AML (Acute Myeloid Leukemia)
Keywords: CAR-T
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: This study is designed as an interventional clinical trial to evaluate the safety and efficacy of anti-CLL1-CD33-NKG2D Bicephali CAR-T cells in patients with relapsed/refractory acute myeloid leukemia (AML). The study will be conducted in a single-arm design, where all participants will receive the experimental treatment. There will be no comparison group or placebo arm.
  Participants in the study will undergo apheresis, a procedure to collect their T cells, which will then be genetically modified to express the anti-CLL1-CD33-NKG2D receptors. After the modification process, these CAR-T cells will be infused back into the patient to target and eliminate AML cells.
  This trial will assess the following key components: Safety and Efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): This arm of the study involves the administration of anti-CLL1-CD33-NKG2D Bicephali CAR-T cells to patients with relapsed/refractory acute myeloid leukemia (AML). Patients will undergo apheresis to collect their T cells, which will then be genetically modified in the laboratory to express the anti-CLL1, CD33, and NKG2D receptors. The modified CAR-T cells will be reinfused into the patient to target and eliminate AML cells. This experimental treatment aims to evaluate the safety, efficacy, and immune response associated with this novel CAR-T therapy.
  Key endpoints include overall survival, progression-free survival, and response rates (such as complete remission or partial remission). Participants will be closely monitored for potential side effects, including cytokine release syndrome (CRS) and neurological toxicity, which are known risks of CAR-T cell therapy.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — This arm of the study involves the administration of anti-CLL1-CD33-NKG2D Bicephali CAR-T cells to patients with relapsed/refractory acute myeloid leukemia (AML). Patients will undergo apheresis to collect their T cells, which will then be genetically modified in the laboratory to express the anti-CLL1, CD33, and NKG2D receptors. The modified CAR-T cells will be reinfused into the patient to target and eliminate AML cells. This experimental treatment aims to evaluate the safety, efficacy, and immune response associated with this novel CAR-T therapy.
  Key endpoints include overall survival, progression-free survival, and response rates (such as complete remission or partial remission). Participants will be closely monitored for potential side effects, including cytokine release syndrome (CRS) and neurological toxicity, which are known risks of CAR-T cell therapy.
  Other Names: anti-CLL1-CD33-NKG2D Bicephali CAR-T cells

SUMMARY:
This study is a clinical trial designed to evaluate the safety and efficacy of a new type of CAR-T cell therapy for patients with relapsed/refractory acute myeloid leukemia (AML). The treatment involves modifying the patient's own T cells to target and eliminate leukemia cells more effectively. This is a cutting-edge therapy using anti-CLL1-CD33-NKG2D Bicephali CAR-T cells.

The primary goal of this study is to determine whether this treatment can improve survival and reduce the symptoms of AML in patients whose disease has not responded to standard treatments. Participants will be closely monitored for side effects and the overall effectiveness of the treatment.

Eligibility for this study includes patients who have been diagnosed with relapsed or refractory AML and have not had success with previous therapies. Participation in this study will provide access to an experimental treatment that may offer benefits beyond current treatment options, but also comes with risks.

Patients, their families, and healthcare providers will be provided with full information about the procedure, potential benefits, and risks, and they will have the opportunity to ask questions before deciding whether to participate.

DETAILED DESCRIPTION:
This clinical trial aims to assess the safety and efficacy of a novel CAR-T cell therapy in patients with relapsed/refractory acute myeloid leukemia (AML). The treatment involves the infusion of genetically modified anti-CLL1-CD33-NKG2D Bicephali CAR-T cells, a type of immunotherapy that enhances the body's immune system to target and destroy cancerous leukemia cells. The therapy is designed to specifically target AML cells by utilizing unique markers (CLL1, CD33, and NKG2D) on the surface of the leukemia cells.

Participants in this study will undergo T cell collection, which involves harvesting their own T cells through a procedure known as apheresis. These cells will then be modified in the laboratory to express the specific CAR-T receptors. Once the cells are modified, they will be re-infused back into the patient, with the goal of activating the immune system to fight off the leukemia.

This study will closely monitor adverse effects, including any side effects of the CAR-T therapy, such as cytokine release syndrome (CRS) or neurological effects, which are known risks of CAR-T treatments. Patients will be followed for a designated period to track response rates, including the reduction of leukemia cells, progression-free survival, and overall survival.

Participants will also undergo regular health assessments, including laboratory tests, imaging studies, and routine examinations, to evaluate both the effectiveness of the treatment and potential complications.

Eligibility for this study includes adult patients with relapsed/refractory AML, meaning their disease has returned after previous treatments or has not responded to standard therapies. This trial provides an opportunity for patients who have limited treatment options to receive access to an advanced, experimental treatment that may improve their outcomes.

Patients will be fully informed about the potential risks and benefits of participating in this study, and their participation will be voluntary. Detailed informed consent will be obtained before any study-related procedures are performed.

ELIGIBILITY:
Inclusion Criteria:

Age: Patients must be ≥18 years old. Diagnosis: Confirmed diagnosis of relapsed or refractory acute myeloid leukemia (AML) as per the World Health Organization (WHO) criteria.

Prior Treatment: Must have failed at least one prior line of chemotherapy or targeted therapy.

Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Adequate Organ Function:

Hematologic function: Absolute neutrophil count (ANC) ≥ 1,000/μL, platelet count ≥ 50,000/μL, and hemoglobin ≥ 8 g/dL (without transfusion support).

Renal function: Serum creatinine ≤ 1.5 x upper limit of normal (ULN). Liver function: Total bilirubin ≤ 2 x ULN, AST/ALT ≤ 2.5 x ULN. Informed Consent: The patient must be willing and able to provide written informed consent to participate in the study.

Eligible for Apheresis: Patients must be able to undergo the apheresis procedure to collect T cells for CAR-T cell modification.

Exclusion Criteria:

Active Central Nervous System (CNS) Leukemia: Presence of active leukemia in the CNS.

Pregnancy or Breastfeeding: Female patients who are pregnant or breastfeeding. Severe Active Infections: Active and uncontrolled infections, including HIV, hepatitis B or C, or any other severe systemic infections.

Other Malignancies: History of another malignancy (except for treated, localized cancers such as basal cell carcinoma) within the past 5 years.

Autoimmune Diseases: Active autoimmune diseases requiring systemic immunosuppressive therapy.

History of Severe Cytokine Release Syndrome (CRS): Any history of severe CRS or neurological toxicity following prior CAR-T cell therapy.

Allergy to Apheresis or CAR-T Cell Components: Known hypersensitivity to any of the components involved in the apheresis or CAR-T cell therapy procedure.

Uncontrolled Systemic Disease: Uncontrolled comorbid conditions, such as severe cardiovascular disease, uncontrolled hypertension, or severe pulmonary conditions.

Concurrent Participation in Another Clinical Trial: Participation in another clinical trial for AML or related conditions that may interfere with this study's treatment and outcomes.

Inability to Comply: Inability to comply with study procedures or follow-up requirements as per the investigator's judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete Remission (CR) or Partial Remission (PR) in Patients with Relapsed/Refractory AML Following CAR-T Therapy | The primary outcome will be assessed at 3 months post-treatment for each participant, with additional follow-up assessments at 6 months and 12 months to monitor remission status
  The primary outcome measure is the rate of complete remission (CR) or partial remission (PR) in patients with relapsed or refractory acute myeloid leukemia (AML) following the administration of anti-CLL1-CD33-NKG2D Bicephali CAR-T cells. CR and PR will be defined according to standard hematologic criteria, including complete resolution or reduction of leukemia cell counts and improvement in bone marrow function. This measure will be assessed using bone marrow biopsies and flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital oh Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Confidentiality and Privacy Concerns: The data collected in this study contains sensitive health information about participants. Protecting patient confidentiality and privacy is of utmost importance, and sharing IPD might pose risks to privacy protections.
  Regulatory Compliance: As the study involves the use of experimental treatments (CAR-T therapy), the sharing of IPD must adhere to strict regulatory guidelines and agreements that protect the intellectual property and ensure the appropriate handling of such data.
  Ongoing Data Analysis: The data from this study is still being analyzed for key outcomes. Sharing incomplete or early-stage data could lead to misinterpretation of the results, affecting the scientific integrity of the study.